CLINICAL TRIAL: NCT02945709
Title: Attention Control Treatment for Post Traumatic Stress Disorder
Brief Title: Attention Control Treatment for Post Traumatic Stress Disorder ׂ(PTSD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor Yair Bar-Haim, Tel Aviv University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAUPTSD
Record Dates: First submitted 2016-10-25; First posted 2016-10-26 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: PTSD
Keywords: PTSD; attention training; cognitive bias modification
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Personalized ACT (Experimental): The personalized attention control training (ACT), comprised of six computerized sessions, in purpose of modulate biases in attention for personalized threat stimuli.
  Interventions: Behavioral: Personalized Attention control training (ACT)
- Non personalized ACT (Active Comparator): The Non-personalized attention control training (ACT), comprised of six sessions, in purpose of modulate biases in attention for non-personalized threat stimuli.
  Interventions: Behavioral: Non-personalized Attention control training (ACT)
- Control training (Placebo Comparator): Computerized control training, comprised of six sessions with a variation of the dot-probe task with neutral stimuli
  Interventions: Behavioral: Control training.

INTERVENTIONS:
Behavioral: Personalized Attention control training (ACT) — In this intervention, participants will be trained with a personalized Dot-Probe task. Each participant will perform the task with the set of words that he or she ranked as the most threatening according to a Word Ranking Task.
  Arms: Personalized ACT
Behavioral: Non-personalized Attention control training (ACT) — In this intervention, participants will be trained with the same Dot-Probe task as in the personalized condition, except that the word stimuli will be randomly fit for each participant. It should be noted that 25% out of the words in this condition will be high ranked words according to each patient's word ranking. The aim of this is to enhance similarity to a generic ACT intervention (see Badura-Brack et al., 2015), where there is some degree of exposure to what one may consider "personalized" stimuli (i.e., threat words that were randomly included by the researchers), although it is not deliberately set to idiosyncratic preferences.
  Arms: Non personalized ACT
Behavioral: Control training. — In this intervention, participants will perform a computerized task, similar to the Dot-Probe task. In each trial, one neutral word will be presented at the center of the screen and participants will respond to a probe ('E' or 'f') presented following the removal of the words display. This version does not include the essential ingredients thought to reduce PTSD symptoms in the other dot-probe tasks: exposure to threat content and competition on attentional resources. Thus, this control version provides a control condition for the ACT interventions.
  Arms: Control training

SUMMARY:
The purpose of this study is to explore the efficacy of Attention Control Training for Post Traumatic Stress Disorder (PTSD).

ACT was found to be effective in decreasing attention bias variability and PTSD symptoms in combat veterans (Badura-Brack, et al., 2015). It is now important to continue the examination of ACT's efficacy in additional populations of patients with PTSD. Such extension of treatment to other traumatic experiences raises the question of whether the threatening content of the training material could be personalized for each patient.

DETAILED DESCRIPTION:
The aim of this study is to explore the efficacy of Attention Control Training for Post Traumatic Stress Disorder (PTSD).

ACT was found to be effective in decreasing attention bias variability and PTSD symptoms in combat veterans (Badura-Brack, et al., 2015). It is now important to continue the examination of ACT's efficacy in additional populations of patients with PTSD. Such extension of treatment to other traumatic experiences raises the question of whether the threatening content of the training material could be personalized for each patient.

For this purpose, we will recruit participants that are diagnosed with PTSD and will be randomly assigned to one of three conditions: personalized ACT, non-personalized ACT, or control training We expect that personalized ACT will produce greater reduction in PTSD symptoms relative to a non-personalized ACT, and that both these conditions will be more effective in symptoms reduction than a control condition not designed to affect attention or expose patients to threat stimuli. We also expect the ACT conditions to reduce attention bias variability relative to the control condition.

ELIGIBILITY:
Inclusion Criteria:

Meeting a current diagnosis of Post-Traumatic Stress Disorder (PTSD) according to DSM-V (American Psychiatric Association, 2013);

Exclusion Criteria:

1. A diagnosis of psychotic or bipolar disorders.
2. A diagnosis of a neurological disorder (i.e., epilepsy, brain injury).
3. Suicidal ideation.
4. Drugs or alcohol abuse.
5. Non-fluent Hebrew.
6. A pharmacological treatment that is not stabilized in the past 3 months (a stable treatment will not be a reason for exclusion from the study).
7. Pregnancy. -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
A diagnosis of PTSD and a total score of severity symptoms, as driven from the CAPS-5 interview | 40 minutes
  The Clinician Administered PTSD Scale (CAPS-5), is a structured interview that will be used to make a diagnosis of PTSD according to the DSM-V criteria. This interview is consists of 30 items regarding the frequency and intensity of PTSD symptoms and a total score of severity is been rated (Weathers, Blake, Schnurr, Kaloupek, Marx, & Keane, 2013).

SECONDARY OUTCOMES:
Total score of the PTSD Checklist (PCL-5). | 10 minutes
  The PCL-5, is a 20-item National Center for PTSD Checklist of the Department of Veterans Affairs. Scores can range from 0 to 80, with higher scores reflecting more symptoms of PTSD (Weathers, Litz, Keane, Palmieri, Marx, & Schnurr, 2013).

OTHER OUTCOMES:
Total score of the PHQ-9 | 10 minutes
  The PHQ-9 , us a 10-item scale for depression symptoms.
The CGI/S | 5 minutes
  Severity and improvement scales (CGI-S/I; Guy, 1976) will be used to assess participants global clinical condition. The CGI-S and the CGI-I are single-items, clinician-reported, measure assessing severity and improvement of illness using a 7-point Likert-type scale. The CGI-S/I has good inter-rater reliability and concurrent validity with other measures. This tool is widely used in clinical trials concerning psychopathology treatments and has good sensitivity to clinical change (e.g., Berk et al., 2008; Hedges, Brown, & Shwalb, 2009; Kadouri, Corruble, & Falissard, 2007; Leon et al., 1993).

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, Prof., Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weathers, F., Blake, D., Schnurr, P., Kaloupek, D., Marx, B., & Keane, T., The clinician-administered PTSD scale for DSM-5 (CAPS-5). Interview available from the National Center for PTSD at www. ptsd. va. gov, 2013.
- [Background] American Psychiatric Association, Diagnostic and Statistical Manual of Mental Disorders (DSM-5). American Psychiatric Pub, 2013
- [Background] Badura-Brack AS, Naim R, Ryan TJ, Levy O, Abend R, Khanna MM, McDermott TJ, Pine DS, Bar-Haim Y. Effect of Attention Training on Attention Bias Variability and PTSD Symptoms: Randomized Controlled Trials in Israeli and U.S. Combat Veterans. Am J Psychiatry. 2015 Dec;172(12):1233-41. doi: 10.1176/appi.ajp.2015.14121578. Epub 2015 Jul 24. PMID 26206075
- [Background] Weathers, F., B. Litz, T. Keane, P. Palmieri, B. Marx, & P. Schnurr, The PTSD Checklist for DSM-5 (PCL-5). Scale available from the National Center for PTSD at www. ptsd. va. gov, 2013.